CLINICAL TRIAL: NCT07349433
Title: Study on 3D-Printed Artificial Airway Fixation Device for Obese Patients: A Randomized Controlled Trial
Brief Title: 3D-Printed Artificial Airway Fixation Device for Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HLXJSXYW-2024-04
Record Dates: First submitted 2025-09-12; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Artificial Airway Management; Obesity &Amp; Overweight
Keywords: 3D Printing; Personalized Fixation Device; Artificial Airway; Endotracheal Intubation; Obesity; Critical Care; Unplanned Extubation; Tube Displacement
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3D-Printed Personalized Fixation Device (Experimental): This arm uses a personalized artificial airway fixation device for obese patients, developed with 3D printing technology, to secure the endotracheal tube.
  Interventions: Device: 3D-Printed Personalized Artificial Airway Fixation Device
- Conventional Fixation Methods (Active Comparator): For Orotracheally Intubated Patients: The standard method involves passing the endotracheal tube through a conventional fixer, tightening the screw cap, and fastening a strap around the neck.
  Interventions: Other: Conventional Fixation Methods

INTERVENTIONS:
Device: 3D-Printed Personalized Artificial Airway Fixation Device — This study uses a personalized artificial airway fixation device for obese patients, developed with 3D printing technology, to secure the endotracheal tube.For Orotracheally Intubated Patients: A fixation device is personalized based on the patient's head and facial contour data. The device is integrally printed with medical-grade silicone-like soft and hard resin, featuring a soft skin-friendly inner side, a rigid movable dual-track structural design, and antimicrobial material on the inner wall.
  Arms: 3D-Printed Personalized Fixation Device
Other: Conventional Fixation Methods — For Orotracheally Intubated Patients: The standard method involves passing the endotracheal tube through a conventional fixer, tightening the screw cap, and fastening a strap around the neck.
  Arms: Conventional Fixation Methods

SUMMARY:
This study is looking for a better way to secure breathing tubes for obese patients who need them. For patients with obesity, a short neck and extra tissue can make it difficult to keep a breathing tube in the correct position. When a tube moves, it can cause serious problems.

Researchers want to compare a new, personalized breathing tube holder with the standard methods currently used.

Participants in this study will be randomly assigned to one of two groups: The Intervention Group will use a new tube holder made with a 3D printer. This holder is custom-designed to fit the specific shape of the patient's face. The Control Group will use the standard methods to secure the breathing tube, such as a conventional holder or medical tape.

Researchers will check things like how well the tube stays in place, the condition of the patient's skin around the mouth, and the comfort of the patient. The goal is to see if the new 3D-printed device is safer, more secure, and more comfortable for obese patients with a breathing tube. The study will include 66 adult patients who are obese and require a breathing tube.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years.
* Meets indications for endotracheal intubation.
* Body Mass Index (BMI) ≥28 kg/m².
* Intact skin around the mouth, cheeks, and neck without lesions before endotracheal intubation.
* Estimated intubation time >12 hours.
* The patient or their family understands and voluntarily participates in this study, and signs the informed consent form.

Exclusion Criteria:

* Patients with a history of psychiatric diagnosis.
* Patients with laryngeal injury.
* Patients with oral diseases or facial skin damage.
* Patients who have undergone intubation more than once during the current hospitalization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2024-07-09 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Endotracheal Tube Displacement or Dislodgement Grade | From intubation through extubation, an average of 7 days.
  The stability of the endotracheal tube is assessed using a 5-point grading scale.
  Grade 1: No displacement. Grade 2: Mild displacement (change of <1 cm). Grade 3: Moderate displacement (change of 1-2 cm). Grade 4: Severe displacement (change of >2 cm). Grade 5: Unplanned extubation (tube is completely dislodged).
Local Skin Integrity | Daily from intubation through extubation, up to 14 days.
  The contact area was inspected daily and recorded for skin irritation or allergic reaction, categorized as "Yes" or "No".
Airway Management Safety Indicators | Average of measurements taken during each oral care procedure from intubation through extubation (an average of 7 days)
  Safety indicators are measured during each nursing procedure (oral care and replacement of the fixation device), including:
  ①Irritative Cough Duration: The duration (in seconds) of a patient's continuous coughing or choking is recorded.
  ②Heart Rate and SpO₂ Fluctuation: Heart rate (beats/minute) and peripheral oxygen saturation (SpO₂) are monitored and recorded before and after each procedure to assess changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
All de-identified individual participant data collected during the study will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The de-identified individual participant data will be publicly shared within 6 months after the first publication of the main research results. The data will remain available for a minimum of 5 years.
Access Criteria: Data will be made available for use by the scientific research community. Access will be provided through a data application and sharing mechanism via the ResMan platform. All shared data will be de-identified to protect participant privacy .
URL: http://www.medresman.org.cn